CLINICAL TRIAL: NCT07148713
Title: Pilot of a CGM-Augmented Food Is Medicine Intervention
Brief Title: Pilot of Continuous Glucose Monitor-Augmented Food Is Medicine
Acronym: ALIGN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-2950; 100001649496 (Other Grant/Funding Number: American Heart Association (AHA))
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-09

CONDITIONS: Nutrition; Type 2 Diabetes; T2DM; T2DM (Type 2 Diabetes Mellitus); Diabetes Education; Diabetes Type 2; Diabetes Mellitis
Keywords: Diabetes; T2DM; Nutrition; Food is Medicine; Continuous glucose monitor; Type 2 Diabetes; Food insecurity; Nutrition insecurity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in the intervention arm will be blinded during Week 0 (Baseline) and Week 12 of the Intervention Phase for a period of 10-14 days to outcome assessments from the CGM wear.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): CGM-Augmented FIM
  Interventions: Behavioral: CGM-Augmented FIM
- Comparator (Active Comparator): FIM only
  Interventions: Behavioral: FIM only

INTERVENTIONS:
Behavioral: CGM-Augmented FIM — The intervention arm will receive electronic healthy foods vouchers and unblinded, real-time CGM sensors for 16-weeks, in addition to individualized nutrition counseling with a registered dietician for 5-8 sessions (all participants will attend 5 sessions, with up to three additional sessions scheduled as needed based a set of a-priori decision rules).
  Arms: Intervention
Behavioral: FIM only — The comparator arm will receive electronic healthy foods vouchers and healthy eating resources and self-directed nutrition education. This group will not receive unblinded CGM sensors or any nutrition counseling for the first 12 weeks. This group will receive 30-days of unblinded CGM sensors to use in the extension phase only.
  Arms: Comparator

SUMMARY:
This study is designed to test the feasibility and preliminary efficacy of a continuous glucose monitor (CGM)-augmented food is medicine (FIM) intervention for adults with type 2 diabetes and nutrition or food insecurity. This study will learn if a FIM intervention ("intervention") that includes access to real-time CGM and nutrition counseling can increase engagement, improve glycemic management, and support healthy eating in this population, compared to the FIM intervention alone ("comparator").

At the study baseline, participants will be randomized to either the intervention or the comparator arm for 16 weeks. The intervention will occur during the first 12 weeks (phase 1: intervention phase) and will be compared to a standard FIM approach without CGM or counseling. Phase 2 (extension phase) will last 4 weeks and will consist of all participants in the intervention and comparator arm receiving both FIM and CGM for self-directed use. The study will also explore participant experiences through a series of semi-structured interviews with a subset of randomly selected participants to identify opportunities for scaling the intervention to a broader population.

DETAILED DESCRIPTION:
This study is designed to test the feasibility and preliminary efficacy of a CGM-augmented FIM intervention for adults with type 2 diabetes and nutrition or food insecurity. The study will enroll adults with type 2 diabetes not using insulin/secretagogues or CGM to be randomized 1:1 to the CGM-augmented FIM intervention (intervention arm) or a standard FIM intervention (comparator arm) for 12 weeks. All participants (N=60) will wear blinded CGM for 10 to 14-days at baseline and at week 12, and complete two random 24-hour dietary recalls during each blinded CGM wear-time. Participants in the intervention arm will wear real-time CGM for the duration of the 12-week intervention and receive a series of structured counseling sessions with a registered dietician. Following the 12-week intervention, all participants will receive both FIM intervention and wear real-time CGM for a 4-week extension phase. FIM intervention will be provided in the form of electronic healthy food vouchers.

At the 12-week and 16-week timepoints, participants will provide outcome data including blinded CGM data, hemoglobin A1c, dietary intake, and other patient-reported outcomes and feedback on their experience using questionnaires. After study completion, a subset of sampled participants will be invited to complete a semi-structured interview regarding their experience with the study. Participants in the intervention group will be invited after the completion of the intervention (beginning week 13) and participants in the comparator group will be invited to interview after completion of the entire study (beginning week 17). The primary outcomes measuring study feasibility and acceptability will collect data related to CGM and FIM use, including overall retention and phase completion, CGM wear-time, use of food subsidy, completion of meal logs, and satisfaction for the intervention. The primary outcomes measuring efficacy will collect diabetes outcomes, glycemic management, and a suite of patient-reported outcomes. Quantitative and qualitative results will be used to improve the intervention prior to rollout of a subsequent multicenter, fully powered randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Able to complete study activities in English
* Aged ≥18 years
* Type 2 diabetes as defined by self-report and confirmed by ICD-10 codes

  * Chart review will be conducted by the study team and a diagnosis of type 2 diabetes (E.11.xx) from either the problem list or a diagnosis linked to an encounter will be used as confirmation. Discrepancies in diagnosis codes will be resolved by review of provider notes within the past 3 years.
* HbA1c > 8.0% in the last 12 months via point of care or venous measurement. If there are multiple values, the most recent one will be considered.
* Receiving primary or specialty care within UNC Health as defined by at least one visit with a primary care provider or endocrine provider within the past year
* Indication of a barrier to healthy eating consisting of report of food insecurity (defined as a score greater or equal to 1.0 on the 6-item USDA Food Security Survey Module (FSSM)) and/OR nutrition insecurity (defined as more often than 'Rarely' on the One-Item Gretchen Swanson Nutrition Screener, OR more often than 'Not Very Hard' on the Two-item Nutrition Security Screener (NSS))

  * Any positive screen on the FSSM, Gretchen Swanson Nutrition Screener, or NSS
* No plans to move from the area for at least 4 months
* Willing and able to provide written informed consent and participate in all study activities

Exclusion Criteria:

* Type 1 or other diabetes
* Use of insulin or secretagogues in the preceding 6 months
* Use of CGM in the preceding 6 months
* Inability to use CGM and related technology (e.g., the companion app), including lack of a smartphone that is compatible with Stelo (information on compatible phones available in Appendix 1) or known allergy to adhesive
* Known psychosis or major psychiatric illness that prevents participation with study activities
* Pregnancy or planned pregnancy in the next 4 months-glycemic targets are different for pregnant women compared to non-pregnant women with diabetes and our intervention is designed for non-pregnant glycemic targets
* Participant in diabetes, nutrition, or weight research intervention in last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in percent of Time in Range (TIR) | Baseline at Week 0, Post-intervention at Week 12
  When using the blinded continuous glucose monitors (CGM), the percentage of sensor values between 70-180 mg/dL will be measured using 7-14 days of retrospective data at each time-point. Change in TIR will be calculated across time-points.
Change in percent of Time Below Range (TBR) | Baseline at Week 0, Post-intervention at Week 12
  When using the blinded continuous glucose monitors (CGM), the percentage of sensor values in the hypoglycemic range (<70 mg/dL) will be measured using 7-14 days of retrospective data at each time-point. Change in TBR will be calculated across time-points.
Change in percent of Time Above Range (TAR) | Baseline at Week 0, Post-intervention at Week 12
  When using the blinded continuous glucose monitors (CGM), the percentage of sensor values in the hyperglycemia range (>180 mg/dL) will be measured using 7-14 days of retrospective data at each time-point. Change in TAR will be calculated across time-points.
Glycemic variability | Baseline at Week 0, Post-intervention at Week 12
  When using the blinded continuous glucose monitors (CGM), glycemic variability will be assessed using the coefficient of variation (%CV). Change in %CV will be calculated across time-points.
Change in Hemoglobin A1c (HbA1c) | Baseline at Week 0, Post-intervention at Week 12
  HbA1c (%) reflects average glucose over the past 2-3 months. Value will be assessed by standardized laboratory assay for trial baseline and endpoint.
Change in Healthy Eating Index (HEI) Score based on two 24-hour recalls | Baseline at Week 0, Post-intervention at Week 12, Post-extension at Week 16
  Participants will be contacted to collect two 24-hour dietary recalls per timepoint. Healthy Eating Index (HEI) scores will be calculated based on the recall responses using a scoring system providing cumulative points for participants eating from a select list of healthy food categories. The scores range from 0 to 100. An ideal overall Healthy Eating Index score of 100 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans (DGA).
Change in Mediterranean diet scores | Baseline at Week 0, Post-Intervention at Week 12, Post-extension at Week 16
  Participants will be contacted to collect two 24-hour dietary recalls per timepoint. Mediterranean diet scores will be calculated based on the recall responses using a scoring system providing cumulative points for participants eating a set amount of serving from a select list of healthy food categories. The scores range from 0 to 9. An ideal overall Mediterranean diet score of 9 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans (DGA).
Change in Dietary Approaches to Stop Hypertension (DASH) Scores | Baseline at Week 0, Post-Intervention at Week 12, Post-extension at Week 16
  Participants will be contacted to collect two 24-hour dietary recalls per timepoint. Dietary Approaches to Stop Hypertension (DASH) scores will be calculated based on the recall responses using a scoring system providing cumulative points for participants eating a set amount of serving from a select list of healthy food categories. The scores range from 8 to 40. An ideal overall DASH score of 40 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans (DGA).

SECONDARY OUTCOMES:
Change in food security using the USDA Food Security Survey Module | Baseline at Week 0, Post-intervention at Week 12, Post-extension at Week 16
  Self-reported United States Department of Agriculture (USDA) Household Food Security Survey will be measured using the 6-item short form with a 30-day lookback period. Responses of either "often", "sometimes", and "yes" on the questionnaire are added up to produce a total raw score, which will be used to measure changes across timepoints in the study. A total raw score of 0-1 indicates high or marginal food security, 2-4 indicates low food security, and 5-6 indicates very low food security.
Change in the presence and/or degree of nutrition security from the Two-item Nutrition Security Screener (NSS) | Baseline at Week 0, Post-Intervention at Week 12, Post-extension at Week 16
  Self-reported 2-item Nutrition Security Screener will be measured to assess the presence and/or degree of nutrition security with the following question: "Thinking about the last 12 months, how hard was it for you or your household to regularly get and eat healthy foods?" The scale yields a nutrition security score based on a 5-point Likert scale ranging from "Very Hard" to "Not hard at all". Responses of "Very Hard", "Hard", or "Somewhat Hard" yield the presence of nutrition insecurity.
Change in the summed nutrition barrier score from the Two-item Nutrition Security Screener (NSS) | Baseline at Week 0, Post-Intervention at Week 12, Post-extension at Week 16
  Self-reported 2-item Nutrition Security Screener will be measured to assess sum of reasons of nutrition barriers with the following question: "People have different reasons for eating or not eating healthy foods. Please tell me which, if any, of the following reasons were true for you or your household in the last 12 months." Participants will have 14 choices to choose from indicating their reason(s) for nutrition barriers, with each reason counting as a score of 1. There is no limit on the number of choices. Each reason checked off will be summed for a total score used to compare between the timepoints for changes in nutrition barrier score.
Change in the One-Item Gretchen Swanson Nutrition Screener | Baseline at Week 0, Post-Intervention at Week 12, Post-extension at Week 16
  Self-reported 1-item Gretchen Swanson Nutrition Screener will be measured to assess the participant's needs for support around accessing healthy foods by asking the following question: "In the last 12 months, I worried that the food I was able to eat would hurt my health and well-being." The scale yields a score based on the response rated on a 6-point Likert scale, ranging from Never, Rarely, Sometimes, Often, Always, and Don't know. Responses with "Sometimes", "Often", and "Always" yields a positive screen, indicating a need for support around accessing healthful foods. Responses with "Never", "Rarely", and "Don't know" yields a negative screen to indicate no need for support around accessing healthful foods.
Change in Core Diabetes Distress using the Type 2 Diabetes Distress Assessment System (T2-DDAS) Core Score | Baseline at Week 0, Post-intervention at Week 12, Post-extension at Week 16
  Self-reported core diabetes distress will be measured using the 29-item Type 2 Diabetes Distress Assessment System (T2-DDAS) Core Score. The scale yields a core score that is the average of all core questions (first 8 items) responses rated on a 5-point Likert scale for all 8 items (range 1-5), with higher scores indicating higher distress. A score >= 2.0 is considered clinically significant diabetes distress.
Change in Sources of Diabetes Distress using the Type 2 Diabetes Distress Assessment System (T2-DDAS) Source Scores | Baseline at Week 0, Post-intervention at Week 12, Post-extension at Week 16
  Self-reported sources of diabetes distress will be measured using the 7 source scales of the 29-item Type 2 Diabetes Distress Assessment System (T2-DDAS) source scale. In addition to the core score, the T2-DDAS scale also yields a score for each of 7 source scales based on the average response on all of the remaining items in the 29-item survey. The 7 source scale scores include: Management Demands, Hypoglycemia, Interpersonal issues, Healthcare provider, Shame/Stigma, Long-term Health, and Healthcare Access. Each of these is measured the same way, on the same 5-point Likert scale (range 1-5), with higher scores indicating higher distress. A score >= 2.0 is considered clinically significant diabetes distress for each source.
Changes in the Benefits of Continuous Glucose Monitor (BenCGM) | Baseline at Week 0, Post-intervention at Week 12, Post-extension at Week 16
  Self-reported BenCGM 8-item survey will be measured. The scale yields a score based on the scale mean taken across all items based on a Likert 5-point scale ranging from 1-5, with a choice of 1 being "Strongly Disagree" to a choice of 5 indicating "Strongly Agree." Changes will be calculated between timepoints
Changes in the Burdens of Continuous Glucose Monitor (BurCGM) | Baseline at Week 0, Post-intervention at Week 12, Post-extension at Week 16
  Self-reported BurCGM 8-item survey will be measured. The scale yields a score based on the scale mean taken across all items based on a Likert 5-point scale ranging from 1-5, with a choice of 1 being "Strongly Disagree" to a choice of 5 indicating "Strongly Agree.". Changes will be calculated between timepoints.
Changes in the 10-item Dietary Screener Questionnaire (DSQ) with a lookback of 30 days. | Baseline at Week 0, Post-Intervention at Week 12, Post-extension at Week 16
  The 10-item Dietary Screener Questionnaire (DSQ) is a validated instrument used to self-report fruit and vegetables intake across different various types of foods. Responses to each question will be sorted either as a fruit, vegetable, or both to generate a score based on intake frequency per month, with choices ranging from "Never" to "6 or more times a day" Results will be calculated by converting the response to cup equivalent estimates of average daily dietary intake and compared across study timepoints.
Change in Physical Activity Levels | Baseline at Week 0, Post-intervention at Week 12, Post-extension at Week 16
  A self-reported Previous Day Physical Activity Recall (PDPAR) will be administered in interview calls measuring frequency of activity from the prior day at the time of the call. Information regarding activity type and intensity levels (ranging light, moderate, hard, and very hard) will be asked for every hour of the wake spent awake. Intensity levels will be used to calculate metabolic equivalent task (MET) values corresponding to each level of intensity to evaluate energy expenditure. MET values will be compared against different timepoints of the study and between study arms.
Change in Food Assistance enrollment (SNAP / WIC) in the last 30 days. | Baseline at Week 0, Post-intervention at Week 12
  Participants will self-report the following question: "Have you received federal food assistance through either SNAP or WIC in the past 30 days." Changes in response of either yes or no will be compared between timepoints.
Changes in financial strain, from the American Academy of Family Physicians (AAFP) Social Needs Screening Tool | Baseline at Week 0, Post-intervention at Week 12
  Participants will self-report the following question from the American Academy of Family Physicians (AAFP) Social Needs Screening Tool: "How often does this describe you? I don't have money to pay my bills (including food, housing, medical care or heating). Never / Rarely / Sometimes / Often / Always" Responses of "Sometimes", "Often", and "Always" yield a positive screen, with a response of "Never" and "Rarely" yielding a negative screen. Scores will be compared between timepoints.
Change in General Health Status | Baseline at Week 0, Post-intervention at Week 12
  Participants will self-report the following question from the General Health Status: "Would you say that in general your health is excellent, very good, good, fair, or poor?" Response will be compared between timepoints.
Change in EuroQol 5 Dimension, 5 Level (EQ-5D-5L) | Baseline at Week 0, Post-intervention at Week 12
  The EuroQol 5 Dimension, 5 Level (EQ-5D-5L) is a self-reported questionnaire that measures general health status in the realms of mobility, self-care, usual activities, pain discomfort, and anxiety/depression. Responses to the 5 questions are based on a Likert 5-point scale measuring severity of problem, with 1 indicating no problems and 5 indicating severe problems. Responses for each question will be concatenated to a 5-digit state in order of mobility, self-care, usual activities, pain discomfort, and anxiety/depression, and then converted to an index score between 0-1. A higher score indicates greater quality of life. Index scores will be compared between timepoints .
Change in overall health status in the EuroQol 5 Dimensions, 5 Level (EQ-5D-5L) | Baseline at Week 0, Post-intervention at Week 12
  The EuroQol 5 Dimension, 5 Level (EQ-5D-5L) is a self-reported questionnaire that measures general health status in the realms of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In the end of the questionnaire, there is a visual analog scale measuring overall health status with the prompt: "We would like to know how good or bad your health is TODAY". Participants will slide the scale to indicate a number ranging from 0 being "The worst health you can imagine" to 100 being "The best health you can imagine". Responses to this question will be compared between timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kahkoska, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 6 to 18 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 6 and continuing for 18 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.